CLINICAL TRIAL: NCT03786237
Title: A Phase II, Open Study to Assess Efficacy and Safety of Rigosertib in Patients With Recessive Dystrophic Epidermolysis Bullosa Associated Locally Advanced/Metastatic Squamous Cell Carcinoma
Brief Title: Rigosertib for RDEB-SCC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Prof. Johann Bauer (Other)
Responsible Party: Sponsor-Investigator, Prof. Johann Bauer, Head of Department of Dermatology, Salzburger Landeskliniken
Organization: Salzburger Landeskliniken (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Rigosertib 5.0
Record Dates: First submitted 2018-11-14; First posted 2018-12-24 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Epidermolysis Bullosa Dystrophica; Squamous Cell Carcinoma
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica; Carcinoma, Squamous Cell | interventions — ON 01910

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Oral Capsules / Intravenous (Experimental)
  Interventions: Drug: Rigosertib Oral Capsules / Rigosertib Intravenous

INTERVENTIONS:
Drug: Rigosertib Oral Capsules / Rigosertib Intravenous — Patients will take Rigosertib either as oral capsules or will get intravenous infusions depending on the needs of the patients.
  Oral Capsules:
  Patients will take oral Rigosertib continuously for a total of three weeks, every four week cycle (three weeks on, one week off drug) for up to 13 cycles. Patients will take 560 mg of oral Rigosertib (ie, 2 capsules of 280 mg) in the morning and in the afternoon, total of 1120mg/day.
  Intravenous Infusions:
  For IV treatment Rigosertib 1800 mg/24 hr is diluted in 0.9% sodium chloride for injection just prior to dosing and is administered as a 72-hr CIV infusion on days 1, 2, and 3 of a 2-week cycle for the first eight 2-week cycles, then on days 1, 2, and 3 of a 4-week cycle thereafter.

SUMMARY:
Epidermolysis bullosa (EB) is a heritable skin disease characterized by marked fragility of epithelialized tissue with blistering in skin and mucous membranes following the slightest mechanical trauma. Eighty percent of all patients suffering from recessive dystrophic EB (RDEB), a subtype originating from mutations in the COL7A1 gene, develop squamous cell carcinoma (SCC). In RDEB patients SCC presents early (most patients are in their 20s or 30s) and shows a highly aggressive metastatic course which often leads to premature death at this young age.

In light of scarce data on the efficacy and safety of systemic treatment regimens for advanced SCC, the investigators propose to perform a small, "first in EB " trial of an experimental drug called rigosertib for the treatment of EB cancer. The trial will be conducted in two study centres, in London and Salzburg, and will last approximately 2.5 years with each patient recruited being in the study for 1 year. The drug is a polo-like kinase inhibitor interfering with different molecular pathways that are essential for cancer cell growth. Rigosertib was developed by Onconova Therapeutics and is currently tested in several clinical trials for a number of other cancers including myelodysplastic syndrome (a cancer of the blood). The investigators have identified that rigosertib most selectively kills EB cancer cells in vitro while leaving normal EB skin cells unaffected. This project will evaluate whether rigosertib is capable of inducing an anti-cancer response in EB patients and whether the drug is well-tolerated. Mechanisms of molecular targeting of squamous cancer cells by rigosertib will further be investigated in EB patients, also aiming at the identification of biomarkers that may allow the predictive identification of best responders.

ELIGIBILITY:
Inclusion Criteria:

1. 18-79 years of age;
2. Diagnosis of unresectable, locally advanced or metastatic SCC confirmed prior to the Screening Visit.
3. Failure to respond to RDEB SCC standard of care, such as surgical excision, radiotherapy or conventional cytotoxic chemotherapy with e.g. platin derivates (i.e.

   cisplatin or carboplatin), 5-fluorouracil, bleomycin, methotrexate, adriamycin, taxanes, gemcitabine or ifosfamide alone or in combination or failure to respond to previous alternative biologic treatments such as epidermal growth factor inhibitors (like cetuximab and panitumumab) or immune checkpoint (programmed cell death

   1) inhibitors (such as nivolumab, pembrolizumab, cemiplimab). For recent guidelines on standard of care for RDEB SCC and non EB-SCC please see Mellerio et al., 2016; Stratigos et al., 2015 and Kim et al., 2018.
4. Is not currently receiving any other cancer therapy.
5. Measurable disease based on Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
6. Patient (or patient's legally authorized representative) must have signed an informed

Exclusion Criteria

1. Response to standard of care.
2. Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure or unstable angina pectoris.
3. Active systemic infection not adequately responding to appropriate therapy.
4. Total bilirubin ≥ 1.5 mg/dL (≥5.3 mg/dL in patients if related to hemolysis or Gilbert's disease).
5. Alanine transaminase (ALT)/aspartate transaminase (AST) ≥ 2.5 x upper limit of normal (ULN).
6. Serum creatinine ≥2 .0 mg/dL or eGFR (estimated Glomerular Filtration Rate) <60mL/min.
7. White blood cell count ≤ 2000/μl, neutrophils ≤ 1500/μL, platelets ≤ 100 x103/μL, hemoglobin ≤ 7.9 g/dL.
8. Known active HIV, hepatitis B or hepatitis C, where active is defined as follows: a. HIV or Hepatitis C - presence of viral load; b. Hepatitis B - antigen positive
9. Uncorrected hyponatremia (defined as serum sodium value of <125 mmol/L).
10. Male patients with partners of child-bearing potential who are unwilling to use male contraception (condom) throughout the study, up to and including the 30-day nontreatment follow-up period.
11. Female subjects: pregnant or lactating women and all women physiologically capable of becoming pregnant (i.e. women of childbearing potential) UNLESS they are willing to use one or more highly effective and reliable methods of contraception with a Pearl index ≤1 including combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral or intravaginal or transdermal); progestogen-only hormonal contraception associated with inhibition of ovulation (oral or injectable or implantable); an intrauterine device (IUD); an intrauterine hormone-releasing system ( IUS); bilateral tubal occlusion; vasectomised partner (provided that partner is the sole sexual partner of the WOCBP trial participant and that the vasectomised partner has received medical assessment of the surgical success) or sexual abstinence (The reliability of sexuality abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject). Reliable contraception should be maintained throughout the study. A pregnancy test in serum will be performed at screening in all women of childbearing potential, and in urine at all visits. Any postmenopausal women (physiologic menopause defined as "12 consecutive months of amenorrhea") or women permanently sterilized (e.g. tubal occlusion, hysterectomy or bilateral salpingectomy) will not be required to undergo pregnancy test.
12. Uncontrolled hypertension. (i.e.. systolic blood pressure greater than or equal to 140mmHg and diastolic blood pressure greater than or equal to 90mmHg despite intake of ≥ 3 antihypertensive medications with complementary mechanisms of action (a diuretic should be 1 component); (Whelton et al., 2018).
13. Patient is currently participating and receiving study therapy or systemic therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
14. Psychiatric illness or social situation that would limit the patient's ability to tolerate and/or comply with study requirements.
15. Patients (or parents in case of paediatric subject) unlikely to comply with the study protocol or unable to understand the nature and scope of the study or the possible benefits or unwanted effects of the study procedures and treatments.
16. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.
17. Known hypersensitivity reaction to any of the components of study treatment.
18. Presence of clinically significant ECG abnormalities based on the inverstigator´s criteria.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Objective Response Rate (ORR) | 1 year
  The primary (efficacy) objective of this trial is to determine the Objective Response Rate (ORR) of therapy with Rigosertib in RDEB patients with locally advanced/metastatic squamous cell carcinoma of the skin using Response Criteria in Solid Tumors Version 1.1 (RECIST1.1) per site assessment up to 52 weeks by CT/MR Scan.
Number of Treatment-related adverse events | 1 year
  Safety will be evaluated for all treated patients, who receive at least one dose of Rigosertib, using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0 (http://ctep.cancer.gov). Safety assessments will be based on number of treatment related adverse events per grade.

SECONDARY OUTCOMES:
Evaluation of quality of life using the "Quality of life in Epidermolysis bullosa questionnaire (QOLEB)" | 1 year
  Assess impact on quality of life using an Epidermolysis bullosa (EB) specific questionnaire developed and published by Murrell et al.2009. Total score is reported (range 0-75; 0 means EB has no affect on ones life, the higher the score the more affect and annoyance/handicap)
Rate of presence or absence of cancer specific biomarkers | 1 year
  Fixed tissue will be assessed using immuno-histochemistry with antibodies raised against phosphorylated AKT (p473 Akt), phosphorylated C-RAF (p-S338 RAF), phosphorylated ERK and cleaved caspase.

CONTACTS AND LOCATIONS:
Overall Officials: Johann W Bauer, Prof., MD, Principal Investigator — Department of Dermatology, Paracelsus Medical University, Salzburger Landeskliniken
Locations (1):
- EB House Austria/Dept. of Dermatology University Hospital, Salzburg, Salzburg, Austria

IPD SHARING:
Plan to Share IPD: Undecided